CLINICAL TRIAL: NCT05621733
Title: A Post Marketing Surveillance of Jakavi® (Ruxolitinib) in Patients With Steroid-Refractory Graft-versus-Host Disease (SR-GvHD) in Korea
Brief Title: A PMS of Jakavi® in Patients With Steroid-Refractory Graft-versus-Host Disease (SR-GvHD) in Korea
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CINC424C2415
Record Dates: First submitted 2022-11-10; First posted 2022-11-18 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Graft-versus-Host Disease
Keywords: Graft-versus-Host disease; GvHD; NIS; Korea; ruxolitinib; Jakavi
MeSH Terms: conditions — Graft vs Host Disease | interventions — ruxolitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- ruxolitinib: Patients currently receiving or going to receive Jakavi® treatment according to locally approved label
  Interventions: Other: ruxolitinib

INTERVENTIONS:
Other: ruxolitinib — Prospective observational study. There is no treatment allocation. Patients prescribed with ruxolitinib in the commercial setting are eligible to enroll into this study.
  Other Names: Jakavi

SUMMARY:
This study is a prospective, open-label, multi-center, non-comparative, observational study to assess safety and effectiveness of Jakavi® (ruxolitinib) in the real-world clinical setting in Korean Graft-versus-Host disease (GvHD) patients

DETAILED DESCRIPTION:
The dosage and duration of treatment may be considered and decided by the investigator in accordance with prescribing information of Jakavi®. All participants who receive at least one dose of the drug and are in the follow-up assessment or early discontinuation (withdrawal) will be the safety population. This study will enroll patients who are newly starting Jakavi® and patients who have been taking Jakavi® prior to study participation. Considering the current clinical practice, a 24 weeks follow-up period of ruxolitinib treatment is needed to assess the safety and the durable effectiveness of the treatment. Mandatory additional safety monitoring will be conducted following the last dose of the treatment for further AE assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who diagnosed with GvHD and currently receiving or going to receive Jakavi® treatment according to locally approved label
2. Patients who are willing to provide written informed consent prior to study enrollment

Exclusion Criteria:

1. Patients under 12 years old
2. Patients with contraindication according to locally approved label of Jakavi®
3. Patients who receive or are going to receive any investigational medicine during the observation period.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are going to receive Jakavi® for the first time or those who are currently taking Jakavi® per clinical judgment
Sampling Method: Non-Probability Sample
Enrollment: 127 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2026-05-09 (Estimated); Study Completion 2026-05-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with an AE/ ADR | Up to 24 weeks
  Proportion of patients with an adverse event (AE)/ adverse drug reaction (ADR) will be provided
Proportion of patients with a SAE/ SADR | Up to 24 weeks
  Proportion of patients with a serious AE (SAE)/ serious ADR (SADR) will be provided
Proportion of patients with an UAE/ UADR | Up to 24 weeks
  Proportion of patients with an unexpected AE (UAE)/ unexpected ADR (UADR) will be provided
Proportion of patients with a SUAE/ SUADR | Up to 24 weeks
  Proportion of patients with a serious unexpected AE (SUAE)/ serious unexpected ADR (SUADR) will be provided

SECONDARY OUTCOMES:
Overall response rate (ORR) | Week 4 and Week 24
  ORR will be analyzed to the proportion of all participants demonstrating complete response (CR) or partial response (PR).
Treatment failure rate | Week 4 and Week 24
  Treatment failure will be analyzed to the proportion of all participants demonstrating lack of response except for CR or PR.
Death rate | Week 4 and Week 24
  Death rate will be provided
Percentage change in CBC | Baseline and Week 24
  Percentage change in CBC (hemoglobin, hematocrit, platelets, white blood cell (WBC) counts) will be provided

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- South Korea (8):
  - Novartis Investigative Site, Daegu, Dalseo gu
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Seoul, Seocho gu
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Jeollanam
  - Novartis Investigative Site, Jinju
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Taegu

IPD SHARING:
Plan to Share IPD: No